CLINICAL TRIAL: NCT04583488
Title: A Phase I Study of Intraperitoneal Docetaxel in Combination With 5-Fluorouracil, Leucovorin, and Oxaliplatin (mFOLFOX6) for Gastric Cancer Patients With Peritoneal Carcinomatosis
Brief Title: Intraperitoneal Docetaxel in Combination With mFOLFOX6 for Gastric Cancer Patients With Peritoneal Carcinomatosis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: PI left institution
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00162730
Record Dates: First submitted 2020-10-05; First posted 2020-10-12 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Peritoneal Carcinomatosis
Keywords: gastric cancer; Peritoneal Surface Malignancies
MeSH Terms: conditions — Peritoneal Neoplasms; Stomach Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intraperitoneal docetaxel (Experimental): Participants will receive intraperitoneal docetaxel combined with the standard of care. A standard 3 + 3 dose escalation design will be used according to the dose escalation plan.
  Interventions: Drug: Intraperitoneal docetaxel

INTERVENTIONS:
Drug: Intraperitoneal docetaxel — Up to 3 dose levels of intraperitoneal docetaxel will be studied (25mg/m2, 35 mg/m2, 45 mg/m2).
  Other Names: Taxotere

SUMMARY:
This is a single-center, open-label, non-randomized, uncontrolled Phase 1 study of intraperitoneal docetaxel in combination with systemic mFOLFOX6 for patients who have gastric cancer with gross peritoneal carcinomatosis (GC-PC).

DETAILED DESCRIPTION:
Gastric cancer (GC) is one of the leading causes of cancer-related deaths in the United States and has a five-year survival of 40% after surgical resection. Metastatic gastric cancer has an even poorer prognosis and most patients die within the first year of diagnosis. Most patients are diagnosed in advanced stages of the disease due to non-specific or lack of symptomatology and treatment options are then limited to systemic chemotherapy. The peritoneum is the most frequent site of metastasis as well as cancer recurrence. Peritoneal Carcinomatosis (PC) results in adverse clinical sequelae and is ultimately responsible for 60% of all gastric cancer-related deaths. While visceral metastases originating from primary gastric cancer are relatively chemosensitive, peritoneal carcinomatosis is particularly challenging to treat because of inadequate drug delivery from systemic circulation. The primary purpose of this trial is to determine the safety of administering intraperitoneal docetaxel in conjunction with the standard of care treatment regimen of intravenous mFOLFOX6 (5-Fluorouracil, leucovorin, and oxaliplatin) in patients with primary gastric cancer with gross peritoneal carcinomatosis.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically-confirmed GC-PC by diagnostic laparoscopy who have not undergone chemotherapy for metastatic/recurrent disease.
* Be willing and able to provide written informed consent/assent for the trial.
* Be ≥ 18 years of age on day of signing informed consent.
* Not have distant metastases as ruled out by an initial imaging (e.g. CT Chest/Abdomen/Pelvis with contrast), positron emission tomography (PET scan). Any metastasis in distant organs other than the peritoneum will exclude the patient from this study.
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale at study entry.
* Demonstrate adequate organ function. All screening labs should be performed within 7 days prior to protocol therapy.
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
* Willingness to undergo intraperitoneal port placement

Exclusion Criteria:

* Has gastric cancer involving the distal esophagus above the gastroesophageal (GE) junction (Siewart type 1, proximally), or second portion of the duodenum (distally).
* Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
* Has a tumor positive for human epidermal growth factor receptor 2 (HER2) staining.
* Has had prior surgery with dense intra-abdominal adhesions
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has had a prior monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 4 weeks (6 weeks for nitrosureas or mitomycin C) prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
* Has known central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has an active infection requiring antibiotic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has any other medical condition, including mental illness or substance abuse, deemed by the Investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C virus (e.g., Hepatitis C virus RNA [qualitative] is detected).
* Patients receiving any medications or substances that are inhibitors or inducers of Cytochrome P450 3A4 (CYP 3A4) are ineligible. Investigator can change to a similar agent that is a non-CYP3A4 inhibitor/inducer with a washout period of 1 week.
* Patients with known hypersensitivity to any of the components of docetaxel or mFOLFOX6.
* Patients who received pelvic or abdominal radiotherapy.
* Peripheral neuropathy ≥ Grade 2.
* History of allogeneic transplant.
* Any known cardiac abnormalities, in accordance with mFOLFOX6 guidelines.
* Any other condition that would render the patient to be unfit for the trial as deemed by the PI or clinical team.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2024-08-06 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 20 weeks
  To determine the Maximum Tolerated Dose (MTD) of intraperitoneal docetaxel in conjunction with the standard of care treatment regimen of intravenous mFOLFOX6 in patients with primary gastric cancer with gross peritoneal carcinomatosis

SECONDARY OUTCOMES:
Progression-Free Survival | 20 weeks
  Progression-free survival rate at 20 weeks, which is defined as the percentage of patients alive and free of disease progression at 20 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Fabian M Johnston, MD, MHS, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No